CLINICAL TRIAL: NCT05633862
Title: Pharmacokinetics, Safety and Tolerability of Doses of BI 1015550 in Healthy Chinese Male and Female Subjects (Open-label, Parallel Group Design)
Brief Title: A Study in Healthy Chinese People to Test How Different Doses of BI 1015550 Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0024
Record Dates: First submitted 2022-11-22; First posted 2022-12-01 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1015550 9 mg (Experimental): A single film-coated tablet of 9 milligram BI 1015550 taken orally after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550
- BI 1015550 18 mg (Experimental): A single film-coated tablet of 18 milligram BI 1015550 taken orally after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — A single film-coated tablet BI 1015550 taken orally after an overnight fast of at least 10 hours.
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
The main objectives of this trial are to investigate pharmacokinetics, safety and tolerability of BI 1015550 in Chinese healthy male and female subjects following administration of single doses.

ELIGIBILITY:
Inclusion criteria

Chinese subjects will only be included in the trial if they meet the following criteria:

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 28.0 kg/m² (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
5. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. Of note, oral hormonal contraceptives are not considered a highly effective method due to potential drug-drug interactions. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the patient information.

Exclusion criteria

Subjects will not be allowed to participate, if any of the following general criteria apply:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder or any history of suicidal ideation or behaviour)
8. History of relevant orthostatic hypotension, fainting spells, or blackouts. Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomised, uncontrolled, open label, single-dose, parallel-group design trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (4.9) | 29.8 (1.9) | 33.3 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Indian | 0 | 0 | 0
  Chinese | 12 | 12 | 24
  Japanese | 0 | 0 | 0
  Korean | 0 | 0 | 0
  Other Asian | 0 | 0 | 0
  Southeast Asian | 0 | 0 | 0
  Taiwanese | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours following drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were treated with at least one dose of trial and who provided at least one pharmacokinetic (PK) endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol*Hour/Liter
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg
Number analyzed (Participants) | 12 | 12
Nanomol*Hour/Liter | 1780 (19.1) | 3680 (32.6)

2. Primary Outcome: Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1015550 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol/Liter
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg
Number analyzed (Participants) | 12 | 12
Nanomol/Liter | 325 (30.3) | 591 (39.0)

3. Secondary Outcome: Number of Subjects With Any Treatment-emergent Adverse Event (AE)
Description: Number of subjects with any treatment-emergent adverse event (AE).
Time Frame: Up to 7 days.
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg
Number analyzed (Participants) | 12 | 12
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Adverse events: Up to 7 days. All-cause mortality: Up to 14 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Arm/Group | BI 1015550 9 mg | BI 1015550 18 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 9 mg (N=12) | BI 1015550 18 mg (N=12)
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Basophil count increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Urinary occult blood positive (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT05633862/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT05633862/SAP_001.pdf